CLINICAL TRIAL: NCT02742090
Title: A Phase 2 Study to Assess the Safety and Efficacy of TGR-1202 (Umbralisib) in Patients With Chronic Lymphocytic Leukemia (CLL) Who Are Intolerant to Prior BTK or PI3K-Delta Inhibitor Therapy
Brief Title: Evaluate the Efficacy and Safety of TGR-1202 in Participants With Chronic Lymphocytic Leukemia Who Are Intolerant to Prior Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: (Strategic/Business Decision)
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGR-1202-201-CLL
Record Dates: First submitted 2016-04-11; First posted 2016-04-18 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — umbralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Umbralisib (Experimental): Participants received 800 milligrams (mg) of umbralisib, orally, once daily until disease progression, unacceptable toxicity or the end of the study for 60.7 months.
  Interventions: Drug: Umbralisib

INTERVENTIONS:
Drug: Umbralisib — Umbralisib was administered as a tablet(s), orally once daily.
  Other Names: TGR-1202

SUMMARY:
The main objective of this study is to determine the progression free survival of umbralisib in participants who were intolerant to prior BTK (Bruton Tyrosine Kinase) inhibitors (ibrutinib, ACP-196, other) or prior PI3K-delta inhibitors (idelalisib, duvelisib, other).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Chronic Lymphocytic Leukemia (CLL)
* Discontinuation on prior BTK inhibitor or PI3K delta inhibitor due to adverse events within prior 9 months
* Presence of measurable disease

Exclusion Criteria:

* Progression on prior BTK or PI3K delta inhibitor
* Prior treatment with TGR-1202
* Richter's transformation or CLL transformation to aggressive lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mato, MD, Study Chair — University of Pennsylvania Center for CLL
Locations (15):
- United States (15):
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Washington D.C., District of Columbia
  - TG Therapeutics Investigational Trial Site, Fort Myers, Florida
  - TG Therapeutics Investigational Trial Site, St. Petersburg, Florida
  - TG Therapeutics Investigational Trial Site, Kansas City, Missouri
  - TG Therapeutics Investigational Trial Site, Lebanon, New Hampshire
  - TG Therapeutics Investigational Trial Site, Hackensack, New Jersey
  - TG Therapeutics Investigational Trial Site, New Hyde Park, New York
  - TG Therapeutics Investigational Trial Site, New York, New York
  - TG Therapeutics Investigational Trial Site, Rochester, New York
  - TG Therapeutics Investigational Trial Site, Durham, North Carolina
  - TG Therapeutics Investigational Trial Site, Hershey, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Philadelphia, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Nashville, Tennessee
  - TG Therapeutics Investigational Trial Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon study closure or as the study evolves

REFERENCES:
- [Derived] Mato AR, Nabhan C, Barr PM, Ujjani CS, Hill BT, Lamanna N, Skarbnik AP, Howlett C, Pu JJ, Sehgal AR, Strelec LE, Vandegrift A, Fitzpatrick DM, Zent CS, Feldman T, Goy A, Claxton DF, Bachow SH, Kaur G, Svoboda J, Nasta SD, Porter D, Landsburg DJ, Schuster SJ, Cheson BD, Kiselev P, Evens AM. Outcomes of CLL patients treated with sequential kinase inhibitor therapy: a real world experience. Blood. 2016 Nov 3;128(18):2199-2205. doi: 10.1182/blood-2016-05-716977. Epub 2016 Sep 6. PMID 27601462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 participants took part in the study at 15 investigative sites in the United States, from 21 April 2016 to 10 June 2021.
Period: Overall Study
Arm/Group | Umbralisib
Started | 51
Completed | 0
Not Completed | 51
Not completed — Adverse Event | 10
Not completed — Death | 3
Not completed — Disease Progression | 25
Not completed — Investigator's Decision | 1
Not completed — Lost to Follow-up | 1
Not completed — Non-compliance with Study | 1
Not completed — Sponsor Discontinuation of the Study | 5
Not completed — Withdrawal by Subject | 4
Not completed — Reason Not Specified | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least one dose of study treatment.
Groups:
- Umbralisib: Participants received 800 mg of umbralisib, orally, once daily until disease progression, unacceptable toxicity or the end of the study for 60.7 months.
  Umbralisib: Umbralisib was administered as a tablet(s), orally once daily.
Arm/Group | Umbralisib
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3
  White | 48

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: PFS was defined as the interval from Day 1 to the earlier of the first documentation of definitive disease progression (PD) or death from any cause. Participants who had no event (progression or death) were censored at the day of their last adequate disease assessment.
Time Frame: From Day 1 to the earlier of the first documentation of definitive disease progression or death (Up to 61.7 months)
Population: The modified Intent to Treat (mITT) population included all participants who were treated with study drug and provided at least one efficacy assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Umbralisib
Number analyzed (Participants) | 47
months | 19.7 [12.9 to 24.8]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR=percent of participants who achieve complete response (CR), or partial response (PR).
Time Frame: Up to 61.7 months
Population: The mITT population included all participants who were treated with study drug and provided at least one efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Umbralisib
Number analyzed (Participants) | 47
percentage of participants | 34

3. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is defined as a composite endpoint measuring time from Day 1 to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death. Estimates of median TTF was made using Kaplan-Meier methods.
Time Frame: From Day 1 to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death (up to approximately 61.7 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Umbralisib
Number analyzed (Participants) | 47
months | 13.6 [9.4 to 19.0]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR defined as the interval from the first documentation of CR or PR to the earlier of the first documentation of definitive disease progression or death from any cause. Estimates of median DOR was made using Kaplan-Meier methods.
Time Frame: From first documentation of CR or PR till disease progression/death (up to approximately 61.7 months)
Population: The mITT population included all participants who were treated with study drug and provided at least one efficacy assessment. Here, Overall number of participants analyzed signifies those who have documented CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Umbralisib
Number analyzed (Participants) | 16
months | 19.4 [8.4 to NA] — Upper limit of 95% CI was not estimable due to low number of participants.

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE's) as Assessed by Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product. An AE does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE is any AE that occur after first dosing of study medication and through the end of the study or through 30 days after the last dose of study treatment, or is considered treatment-related regardless of the start date of the event, or is present before first dosing of study medication but worsens in intensity or the investigator subsequently considers treatment-related. TEAEs included both serious and non-serious TEAEs.
Time Frame: From first dose of study treatment up to end of study (up to 61.7 months)
Population: The safety population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbralisib
Number analyzed (Participants) | 51
Participants | 51

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to end of study (up to approximately 61.7 months)
Description: The safety population included all participants who received at least one dose of study treatment.
Arm/Group | Umbralisib
All-Cause Mortality (participants affected / at risk) | 3/51
Serious Adverse Events (participants affected / at risk) | 22/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Umbralisib (N=51)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Atrial fibrillation (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 7
Influenza (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Influenza A virus test positive (Investigations) | 1
Platelet count decreased (Investigations) | 1
Transaminases increased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Urticaria (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Umbralisib (N=51)
Anaemia (Blood and lymphatic system disorders) | 7
Leukocytosis (Blood and lymphatic system disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 36
Nausea (Gastrointestinal disorders) | 32
Constipation (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 12
Oedema peripheral (General disorders) | 10
Pyrexia (General disorders) | 7
Upper respiratory tract infection (Infections and infestations) | 9
Contusion (Injury, poisoning and procedural complications) | 11
Aspartate aminotransferase increased (Investigations) | 10
Neutrophil count decreased (Investigations) | 10
Alanine aminotransferase increased (Investigations) | 9
Blood alkaline phosphatase increased (Investigations) | 7
Platelet count decreased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 10
Hypokalaemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Headache (Nervous system disorders) | 14
Dizziness (Nervous system disorders) | 8
Paraesthesia (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 5

LIMITATIONS AND CAVEATS:
Due to sponsor's business decision, the clinical trial was terminated by the sponsor prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is restricted from publication until after the multi-center paper is published.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT02742090/Prot_SAP_000.pdf